CLINICAL TRIAL: NCT03346044
Title: Medtronic's MOSAIC Bioprosthesis Versus Baxter Carpentier-Edwards SAV Porcine Valve: A Longterm Prospective Randomized Clinical Evaluation
Brief Title: Medtronic's MOSAIC Bioprosthesis Versus Baxter Carpentier-Edwards SAV Porcine Valve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Principal Investigator, Michael Jonathan Unsworth-White, Consultant Cardiothoracic Surgeon, University Hospital Plymouth NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1301
Record Dates: First submitted 2017-09-08; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Cardiac Valve Replacement

STUDY DESIGN:
Intervention Model Description: A comparative single centre study of two porcine bioprostheses indicated for the surgical treatment of heart valve diseases. The study will compare two equal sized patient groups using either the Medtronic Mosaic and Carpentier-Edwards SAV bioprostheses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carpentier-Edwards SAV bioprostheses (Active Comparator)
  Interventions: Device: Carpentier-Edwards SAV bioprostheses
- Medtronic Mosaic bioprostheses (Active Comparator)
  Interventions: Device: Medtronic Mosaic bioprostheses

INTERVENTIONS:
Device: Carpentier-Edwards SAV bioprostheses — Performance of these bioprostheses
  Arms: Carpentier-Edwards SAV bioprostheses
Device: Medtronic Mosaic bioprostheses
  Arms: Medtronic Mosaic bioprostheses

SUMMARY:
The study compares the clinical performance of the Mosaic valve with that of the Baxter valve (Carpentier-Edwards) which is widely used throughout the UK and is considered to be the "bench mark".

Specific objectives will be to determine structural failure and valve explantation rates, thromboembolic events and mortality rates for each valve.

Haemodynamic assessments will also be made using echocardiography to measure gradients across the valves and changes in left ventricular function and wall thickness.

DETAILED DESCRIPTION:
The bioprostheses (xenografts) to be used in this study are third generation valves derived from porcine aortic valves. The chief advantage over mechanical prostheses is that they do not require lifelong anticoagulation with warfarin with its attendant risks of haemorrhage if the patient becomes over anticoagulated, or thromboembolism if anticoagulation is inadequate. However their disadvantage is that they are prone to calcification and mechanical failure over time. Because of this, bioprosthetic valves are usually reserved for older patients in whom the chance of repeat surgery is reduced.

The Medtronic Mosaic stented bioprosthesis has been recently introduced. The Mosaic bioprosthesis utilizes Physiological Fixation (root fixation with zero pressure differential across the valve leaflets). This allows valves to maintain their natural leaflet structure and root geometry. The Mosaic bioprosthesis uses the AOA anti-mineralisation treatment. Developed in collaboration with Biomedical Design, Inc., AOA has been shown in multiple animal studies to be an effective treatment in preventing leaflet calcification.

Baxter currently produces the Carpentier Edwards SAV porcine bioprosthesis that has abundant long-term follow-up data and is widely used. Low pressure fixation (less than 1.5mmHg) and anti-mineralisation treatment with FET 80TM are used in its preparation. The stent (which supports the cusps) has been designed to allow for the wider opening angle of the softer leaflets.

These features aim to improve on the haemodynamic performance of earlier generation valves and offer the potential for increased durability. Early results look promising with excellent haemodynamic parameters and remarkably low rates of structural failure.

If zero pressure fixation and anti-mineralisation treatment can be shown to increase the longevity of the bioprosthetic valve, the age criteria for implantation will undoubtedly be lowered allowing a younger cohort of patients to benefit from anticoagulation-free therapy and freedom from associated morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require isolated or combined aortic or mitral valve replacement with or without coronary artery bypass grafting
* Patients requesting anticoagulation-free therapy
* Patients who are able to provide informed consent

Exclusion Criteria:

* Concomitant procedures other than coronary artery bypass grafting
* Presence of illness other than valve disease that would substantially increase the likelihood of death within one year
* Patients unlikely to be available for long term follow-up activities
* Patients indicated for receiving a mechanical prosthesis
* Patients refusing or not able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2001-01-01 (Actual); Primary Completion 2006-02-02 (Actual); Study Completion 2016-01-12 (Actual)

PRIMARY OUTCOMES:
Mortality | 10 years
  Early mortality was defined as death occurring within 30 days of implantation if the patient was discharged from hospital or at any time after implantation if the patient was not discharged from hospital. Hospital-to-hospital transfer was not considered as discharge. Late mortality was defined as all deaths that occurred after 30 days of implant, if the patient was discharged from hospital.
  The reporting of mortality and morbidity follows the guidelines of the Society of Thoracic Surgeons (STS), the American Association of Thoracic Surgeons (AATS) and the European Association for Cardiothoracic Surgery (EACTS). () Edmunds LH, Clark R, Cohn L, et al. Guidelines for Reporting Morbidity and MortalityAfter Cardiac Valvular Operations. Ann Thorac Surg 1996;62:932-5)
Freedom from structural valve deterioration (SVD) | 10 years
  Defined as re-operation and thromboembolic events. Valve-related complications were defined as thromboembolism, structural valve dysfunction, non-structural valve dysfunction and prosthetic valve endocarditis.

SECONDARY OUTCOMES:
Haemodynamic performance (mmHg) | 10 years
  Transvalvular gradients measured in mmHg
Left ventricular (LV) mass regression (grams) | 10 years
  Evidence of left ventricular mass regression measured in grams

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Unsworth-White, BSc FRCS, Principal Investigator — University Hospital Plymouth NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zibdeh O, Bugg I, Patel S, Twine G, Unsworth-White J. Randomized trial of the Carpentier-Edwards supra-annular prosthesis versus the Medtronic Mosaic aortic prosthesis: 10-year results. Eur J Cardiothorac Surg. 2018 Aug 1;54(2):281-287. doi: 10.1093/ejcts/ezx512. PMID 29401266